CLINICAL TRIAL: NCT03189147
Title: BicepsTenodesis vs. Biceps Debridement in Combined Rotator Cuff (RC) Tears and Superior Labral Anterior to Posterior (SLAP) Lesions: A Randomized Trial
Brief Title: BicepsTenodesis vs. Biceps Debridement in Combined RC Tears and SLAP Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low recruitment rate
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00072759
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: SLAP Lesion
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biceps Tenodesis (Experimental): Patients in this group will received biceps tenodesis intervention to address their labral lesion
  Interventions: Procedure: Biceps Tenodesis
- Debridement (Active Comparator): Patients in this group will received debridement intervention to address their labral lesion
  Interventions: Procedure: Debridement

INTERVENTIONS:
Procedure: Biceps Tenodesis — Surgical procedure that is usually performed for the treatment of labral lesions in patients undergoing arthroscopic rotator cuff repair
  Arms: Biceps Tenodesis
Procedure: Debridement — Surgical procedure that is usually performed for the treatment of labral lesions in patients undergoing arthroscopic rotator cuff repair
  Arms: Debridement

SUMMARY:
The appropriate treatment of labral lesions such as SLAP tears in patients undergoing RC tears repair is controversial. Most surgeons are reluctant to repair RC and SLAP tears simultaneously due to the high likelihood of prolonged postoperative immobilization, stiffness and poor clinical outcomes. The current standard care interventions include debridement, biceps tenotomy or tenodesis rather than surgical repair of SLAP tears. Simple debridement is a low cost and time-saving procedure that has the advantage of maintaining the anatomy of the long head of biceps (LHB), a muscle that acts as an active depressor of the head of the humerus in patients with RC tears. Biceps tenotomy is also low cost and time-saving; however, since the LHB is released from its attachment in the shoulder joint, the anatomy is not preserved and results in decreased strength and possible development of a 'Popeye' deformity. Biceps tenodesis has higher costs and time than the other two approaches, but has the advantage of preserving the LHB anatomy and power, and a lower possibility of developing complications. Finally, labral repair has the highest costs and associated surgical time and may lead to increase stiffness after surgery, particularly in patients over 45 years old.

Currently, the standard care of the surgeons involved in this study is to use either debridement or biceps tenodesis to address labral lesions in patients undergoing surgery for their RC tear. Based on the current evidence and current practice in our facility, we aim to compare the efficacy of tenodesis versus debridement in patients with combined RC tear, degenerative labrum (SLAP tears) and a normal biceps tendon.

DETAILED DESCRIPTION:
Rotator cuff (RC) tears are the most common source of shoulder pain, disability and discomfort. In fact, RC disease is the most common cause of shoulder pain seen by physicians. It has been estimated that as many as 40% of patients with shoulder pain may have a RC tear. Previous research has shown that 80% of these patients will experience pain, and 40% of patients will experience tear progression (tear becoming larger, more painful, multiple muscle involvement). Therefore, it is no surprise that a substantial proportion of individuals with RC tears do not receive adequate relief from non-operative treatments (physiotherapy, acupuncture, massage therapy, activity/work modification, cortisone injection), and require surgical repair.

Surgical repair has been challenging in this population, since frequently RC tears are associated with concomitant labral lesions such as SLAP (superior labral anterior-posterior) tears that may increase patients' symptoms. Miller and Savoie studied one hundred patients with full-thickness RC tears and determine that 74% had coexisting intra-articular abnormalities, and labral tears were the most common associated pathology. Gartsman et al reported that 60.5% of patients with full-thickness RC tears had coexisting intraarticular abnormalities, with 25 patients (12.5%) having major abnormalities that required surgery, changed postoperative rehabilitation or impacted the expected end result. Snyder et al. 8 reported that 40% of patients with SLAP lesions had associated full- or partial-thickness RC tears.

The appropriate treatment of labral lesions such as SLAP tears in patients undergoing RC tears repair is controversial. Most surgeons are reluctant to repair RC and SLAP tears simultaneously due to the high likelihood of prolonged postoperative immobilization, stiffness and poor clinical outcomes. Therefore, the current standard care interventions include debridement, biceps tenotomy or tenodesis rather than surgical repair of SLAP tears3. Recently, Oh et al. compared simple debridement, biceps tenotomy, and biceps tenodesis for the patients with concomitant RC tear and labral lesions. All concomitant treatments improved patients' symptoms. Simple biceps debridement had the lowest risk of patients developing a 'Popeye' deformity and preserved forearm supination strength. Biceps tenotomy appeared preferable for patients with definite groove tenderness while biceps tenodesis was indicated for patients with groove tenderness, but who wanted to preserve supination strength. However, this study was compromised by low follow-up (72%) within one year and unbalanced groups (i.e.one group had significantly more males). Abbot et al. determined that patients over the age of 45 years treated with arthroscopic RC repair and SLAP debridement had significantly better function, pain relief, and range of motion than those treated with RC repair and simultaneous SLAP repair. A systematic review in 2011 looked at the current evidence for effectiveness of interventions to treat RC tears, and they found limited evidence favoring debridement compared to anchor replacement and suture repair of Type II SLAP tear. Another systematic review in 2014 revised the published data on the surgical treatment of superior labral injuries in patients aged 40 years, including those with concomitant injuries to the RC and they stated that the cumulative evidence supports labral debridement or biceps tenotomy over labral repair when an associated RC injury is present.

The above studies are contradictory likely because studies were heterogeneous in terms of selection as well as assessment periods and outcome measurements performed. Therefore, the question about best practice to treat labral lesions in patients with concomitant RC tears remains unanswered.

Moreover, in previous studies, surgical time and costing with the different approaches were not considered. Simple debridement is a low cost and time-saving procedure that has the advantage of maintaining the anatomy of the long head of biceps (LHB), a muscle that acts as an active depressor of the head of the humerus in patients with RC tears. Biceps tenotomy is also low cost and time-saving; however, since the LHB is released from its attachment in the shoulder joint, the anatomy is not preserved and results in decreased strength and possible development of a 'Popeye' deformity. Biceps tenodesis has higher costs and time than the other two approaches, but has the advantage of preserving the LHB anatomy and power, and a lower possibility of developing complications. Finally, labral repair has the highest costs and associated surgical time and may lead to increase stiffness after surgery, particularly in patients over 45 years old.

Currently, the standard care of the surgeons involved in this study is to use either debridement or biceps tenodesis to address labral lesions in patients undergoing surgery for their RC tear. Annually, in the Edmonton region, as an estimate from all of the surgeons involved in this study, surgeons perform around 200 of each technique (debridement or biceps tenodesis). Based on the current evidence and current practice in our facility, we aim to compare the efficacy of tenodesis versus debridement in patients with combined RC tear, degenerative labrum (SLAP tears) and a normal biceps tendon.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 35 years of age presenting with a high grade partial-thickness or full-thickness RC tear associated with a degenerative SLAP tear and a normal biceps tendon, confirmed by appropriate imaging, that can be surgically repaired using an arthroscopic approach will be eligible for the study.

Exclusion Criteria:

* Subjects presenting with pulley involvement, high grade full-thickness RC tears (>3cm), biceps pathology, previous surgery to the affected shoulder, history of shoulder dislocation, inflammatory disease, or moderate to severe degenerative glenohumeral arthropathy (Kellgren-Lawrence Grade 3 or 4), major shoulder joint trauma, infection, or avascular necrosis will be excluded. Furthermore, those with psychiatric illness, cognitive impairment, or health conditions that preclude informed consent, life expectancy of less than 1 year, who do not speak/read/understand English, have no fixed address or contact, or are unwilling to complete follow-ups will also be excluded

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) in different time points | Baseline, 2-weeks, 6-weeks, 3-months, 6-months and 12-months
  Pain at rest, sleep and with activity will be measured using an 11-point VAS (0-10), a reliable and valid method of measuring patient-reported pain.

SECONDARY OUTCOMES:
Range of Motion | Baseline, 6-weeks, 3-months, 6-months and 12-months
  Active and passive ROM assessments of shoulder flexion, abduction, external rotation (90° abduction, 90° elbow flexion), and internal rotation (90° abduction, 90° elbow flexion) will be conducted by the research coordinator for both the affected and unaffected shoulder at baseline and only affected arm on follow-ups.

OTHER OUTCOMES:
Shoulder Flexion Strength | Baseline, 6-months and 12-months
  Strength assessments will also be conducted by the research coordinator at baseline and 6- and 12-months. Strength will be measured by using peak values of isometric shoulder flexion, using a hand held dynamometer (microFET3, Hoggan Health Industries Inc., West Jordan, UT).
Shoulder Abduction Strength | Baseline, 6-months and 12-months
  Strength assessments will also be conducted by the research coordinator at baseline and 6-, and 12-months. Strength will be measured by using peak values of isometric shoulder abduction, using a hand held dynamometer (microFET3, Hoggan Health Industries Inc., West Jordan, UT).
Shoulder External Rotation Strength | Baseline, 6-months and 12-months
  Strength assessments will also be conducted by the research coordinator at baseline and 6-, and 12-months. Strength will be measured by using peak values of isometric shoulder external rotation, using a hand held dynamometer (microFET3, Hoggan Health Industries Inc., West Jordan, UT).
Shoulder Internal Rotation Strength | Baseline, 6-months and 12-months
  Strength assessments will also be conducted by the research coordinator at baseline and 6-, and 12-months. Strength will be measured by using peak values of isometric shoulder internal rotation, using a hand held dynamometer (microFET3, Hoggan Health Industries Inc., West Jordan, UT).
Elbow supination Strength | Baseline, 6-months and 12-months
  Strength assessments will also be conducted by the research coordinator at baseline and 6-, and 12-months. Strength will be measured by using peak values of isometric elbow supination, using a hand held dynamometer (microFET3, Hoggan Health Industries Inc., West Jordan, UT).
Western Ontario Rotator Cuff Index Index (WORC) | Baseline, 6-weeks, 3-months, 6-months and 12-months
  The WORC is a 5-part (physical symptoms, sports/recreation, work, lifestyle, emotions), 21-item, disease-specific questionnaire that assesses quality of life in subjects with RC pathology. The WORC has been proven to be a valid, reliable and responsive tool in this population.
Visual analysis of biceps contraction to check for any signs of Popeye Deformity | 2-weeks, 6-weeks, 3-months, 6-months and 12-months
  Signs of popeye deformity will be noted during all follow-ups if any

CONTACTS AND LOCATIONS:
Locations (1):
- Sturgeon Community Hospital, St. Albert, Alberta, Canada